CLINICAL TRIAL: NCT07320534
Title: The Effect of Levofloxacin Prophylaxis on the First Occurrence of Febrile Neutropenia During Induction Chemotherapy in Pediatric Patients With Acute Lymphoblastic Leukemia at Dr. Sardjito Hospital
Brief Title: Levofloxacin Prophylaxis to Prevent First Febrile Neutropenia in Pediatric ALL During Induction Phase
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Dr. Sardjito Hospital, Yogyakarta (Unknown)
Responsible Party: Principal Investigator, Idha Yulandari, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KE/FK/1504/EC/2025
Record Dates: First submitted 2025-09-24; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neutropenic Fever; Acute Lymphoblastic Leukemia
Keywords: Neutropenic Fever; Acute Lymphoblastic Leukemia; Levofloxacin
MeSH Terms: conditions — Febrile Neutropenia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Levofloxacin (Experimental): Receiving oral levofloxacin as infection prophylaxis during the induction phase, with the following dosage:
  * Age < 5 years: 10 mg/kg PO every 12 hours (maximum 250 mg/dose)
  * Age ≥ 5 years: 10 mg/kg PO once daily (maximum 500 mg/day)
  Interventions: Drug: Levofloxacin
- Group B: Placebo (Placebo Comparator): Receiving oral placebo at the same dosage as the treatment group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levofloxacin — younger than 5 years received levofloxacin 10 mg/kg by mouth every 12 hours and patients 5 years and older received 10 mg/kg by mouth once daily (maximum 500 mg/dose)
  Arms: Group A: Levofloxacin
Other: Placebo — Receiving oral placebo at the same dosage as the treatment group.
  Arms: Group B: Placebo

SUMMARY:
The goal of this clinical trial is To evaluate the benefit of levofloxacin prophylaxis in prolonging the median time to first febrile neutropenia in pediatric ALL patients during induction phase. It will also learn about the safety of levofloxacin during induction treatment.

The main questions it aims to answer are:

* Does levofloxacin prophylaxis increase the median time to the first febrile neutropenia episode compared to placebo?
* What are the rates of fever, severe infection, organ-related bacterial infection, and mortality in children receiving levofloxacin compared to placebo?

Researchers will compare oral levofloxacin to a placebo (a look-alike substance with no active drug) to see if levofloxacin is effective in preventing infection during induction chemotherapy.

Participants will:

* Be children aged 1 to 18 years with ALL undergoing induction chemotherapy.
* Be randomly assigned to receive either levofloxacin prophylaxis or placebo during the induction phase.
* Have regular checkups, physical exams, and laboratory tests during induction.
* Be monitored for fever, febrile neutropenia, severe infections, bacterial infections, and mortality.
* Stop prophylaxis once the first febrile neutropenia occurs or induction therapy is completed.

DETAILED DESCRIPTION:
Furthermore, this clinical trial aims to:

* To determine the incidence of fever during the induction phase in pediatric ALL patients receiving levofloxacin prophylaxis compared with placebo.
* To determine the incidence of febrile neutropenia during the induction phase in pediatric ALL patients receiving levofloxacin prophylaxis compared with placebo.
* To determine the incidence of severe infections during the induction phase in pediatric ALL patients receiving levofloxacin prophylaxis compared with placebo.
* To determine the number of organ-related bacterial infections, whether microbiologically confirmed or not, during the induction phase in pediatric ALL patients receiving levofloxacin prophylaxis compared with placebo.
* To determine the mortality rate during the induction phase in pediatric ALL patients receiving levofloxacin prophylaxis compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 1 to 18 years diagnosed with acute lymphoblastic leukemia (ALL).
* Receiving induction phase 1A chemotherapy for ALL using the Indonesian National Childhood ALL Pilot Protocol 2024 Standard Risk; induction phases 1A and 1B chemotherapy using the Indonesian National Childhood ALL Pilot Protocol 2024 High Risk; or induction chemotherapy using the ACT4ALL Protocol 2025 at Dr. Sardjito Hospital.
* No history of allergy to levofloxacin.
* Parents/guardians provide written informed consent.

Exclusion Criteria:

* Death before initiation of chemotherapy.
* Patients with clinically or microbiologically confirmed infection within 72 hours prior to induction chemotherapy who require antibiotics for more than 5 days (to avoid antibiotic therapy as a confounding factor for antibiotic prophylaxis).

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Median time to first febrile neutropenia | First febrile neutropenia up to day 63
  The number of participants with first febrile neutropenia and the median day of occurrence.
Clinical Outcome | First febrile neutropenia up to day 63
  The number of participants who experienced fever, first febrile neutropenia, severe infection, organ-related infection, microbiologically confirmed infection, infection-related mortality

SECONDARY OUTCOMES:
Caused of mortality | up to 12 weeks
  The cause of mortality in the participants.
Patients with positive cultures | up to 12 weeks
  The number of participants who were positive for bacteria or fungi, and the number of participants with antibiotic resistance (resistant to fluoroquinolones, carbapenems, or vancomycin).

OTHER OUTCOMES:
Baseline characteristics of the study groups | Day 1
  Number of participants with each variable:
  Age (only 2 variations)
  * <10 years
  * ≥10 years
  Sex
  * Male
  * Female
  Nutritional Status Categories of Children Aged ≤ 10 Years Based on WHO BMI-for-Age Z-scores (BMI in kg/m^2)
  * Severely wasted
  * Wasted
  * Normal
  * Possible risk of overweight
  * Overweight
  * Obese
  BMI Classification for Children Aged > 10 Years Based on BMI (kg/m^2)
  * Underweight
  * Normal
  * Overweight
  * Obesity
  Leukemia risk group (only 2 variation, using the Indonesia Pilot Protocol 2024)
  * Standard risk
  * High risk

CONTACTS AND LOCATIONS:
Overall Officials: Idha Yulandari, M.D. Pediatric, Principal Investigator — Gadjah Mada University
Locations (1):
- RSUP dr Sardjito, Sleman, DI Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Inform Consent Form
Supporting Information: ICF
Time Frame: 07 October 2025 for 1,5 years
Access Criteria: No data will be shared publicly. Data access will only be provided to qualified researchers upon justified request and with ethics approval.
URL: https://drive.google.com/file/d/1BGYHRI1fgXd5k7X0VABCEte6_RG_YB_O/view?usp=drive_link

REFERENCES:
- [Result] Alexander S, Fisher BT, Gaur AH, Dvorak CC, Villa Luna D, Dang H, Chen L, Green M, Nieder ML, Fisher B, Bailey LC, Wiernikowski J, Sung L; Children's Oncology Group. Effect of Levofloxacin Prophylaxis on Bacteremia in Children With Acute Leukemia or Undergoing Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2018 Sep 11;320(10):995-1004. doi: 10.1001/jama.2018.12512. PMID 30208456
- [Result] Patel B, Noda A, Godbout E, Stevens M, Noda C. Levofloxacin for Antibacterial Prophylaxis in Pediatric Patients With Acute Myeloid Leukemia or Undergoing Hematopoietic Stem Cell Transplantation. J Pediatr Pharmacol Ther. 2020;25(7):629-635. doi: 10.5863/1551-6776-25.7.629. PMID 33041718